CLINICAL TRIAL: NCT03118882
Title: Pilot RCT on Lifestyles Impact on Health Outcomes in the General Population Invited to Mammography and Colorectal Cancer Screening Programmes. (STI.li di VI.ta - Lifestyles) STI.VI.
Brief Title: STI.VI. Study: How to Improve Lifestyles in Screening Contexts
Acronym: STIVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro di Riferimento per l'Epidemiologia e la Prev. Oncologica Piemonte (Other)
Collaborators: Azienda Sanitaria Locale Torino 1 (Unknown)
Responsible Party: Principal Investigator, Nereo Segnan, Director, S.C. Epidemiologia, Screening e Registro Tumori Centre for Cancer Prevention, Principal investigator, Centro di Riferimento per l'Epidemiologia e la Prev. Oncologica Piemonte
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pratica 2008.1405 Prot.1362
Record Dates: First submitted 2017-03-31; First posted 2017-04-18 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Lifestyle Risk Reduction; Weight Changes, Body; Breast Cancer; Colorectal Cancer
Keywords: Breast cancer screening; Colorectal Cancer screening; Primary prevention; Lifestyles; Teachable moment
MeSH Terms: conditions — Risk Reduction Behavior; Body Weight Changes; Breast Neoplasms; Colorectal Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Diet Group (Active Comparator)
  Interventions: Behavioral: Diet group
- Physical activity group (Active Comparator)
  Interventions: Behavioral: Physical activity group
- Physical activity and diet group (Active Comparator)
  Interventions: Behavioral: Physical activity and diet group
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Diet group — A meeting where an expert illustrates the scientific basis of a proper diet. Moreover, clear and practical indications for dietary habits improvement and for suggested food purchase are provided. After having completed the basic module, participants are offered the opportunity of deepening the educational process through an advanced module:hree theoretical and practical cooking meetings (total of 10 hours) held by cooks with an expertise in natural cuisine and by trained dieticians.
  Arms: Diet Group
Behavioral: Physical activity group — A meeting where an expert illustrates the benefits of a constant PA. Moreover, indications are given on sport opportunities and walking groups in the city organised by public authorities. After having completed the basic module, participants are offered the opportunity of deepening the educational process through an advanced module: three theoretical and practical lessons (total of 10 hours) held by expert physical trainers.
  Arms: Physical activity group
Behavioral: Physical activity and diet group — A meeting where the indications given to the previous groups are presented simultaneously. Particular attention is paid to the interaction between the two activities. After having completed the basic module, participants are offered the opportunity of deepening the educational process through an advanced module: four theoretical and practical meetings (total of 12 hours), two lessons focus on diet and two on PA.
  Arms: Physical activity and diet group

SUMMARY:
The main study objective is to determine the feasibility and impact (effectiveness) of intervention models for lifestyle changing (diet and physical activity) on health outcomes. Women 50 to 54-year-old attending the local breast cancer screening and 58-year-old people (both sexes) undergoing colorectal cancer screening are invited to participate in the study. Compliers are randomized into 3 intervention groups (Diet, Physical Activity, and Physical Activity and Diet) and into the 'usual care' Control group. Biological sampling (blood and saliva) is collected from all participants. All participants undergo also anthropometric measurements and fill in a self-administered validated questionnaire on their dietary and physical activity habits. All enrolled subjects receive a booklet with basic information about diet and physical activity. Subjects randomized to the 3 intervention groups are also offered one theoretical and three training courses. The courses are specifically designed for the different interventions proposed and aimed at reinforcing the educational counseling and at supporting behavioral changes.

Follow-up is performed at 8 (intermediate follow-up) and 12-14 (final follow-up) months for repeating anthropometric measurements and questionnaire filling and blood sampling (at the final one).

DETAILED DESCRIPTION:
The study aims to evaluate the effectiveness of intervention models on diet and physical activity.

The study randomizes eligible subjects into four groups: Diet group, Physical Activity group, Physical Activity and Diet group and "Usual Care" control group. To each group a specific intervention is delivered, consisting of counselling, informative material, and dedicated training.

All participants (with the exception of the control group) receive a basic counselling by field experts. Afterwards they are offered an advanced training including more specific and detailed actions.

An information booklet specifically developed for this study is distributed to all participants. The booklet contains general information on primary prevention, based on the most reliable and updated bibliographic sources on diet and physical exercise.

Together with the letter of screening invitation eligible men and women receive the proposal to participate in the STI.VI. study. Participation to screening is not considered a prerequisite for study participation. A direct phone number and e-mail address are given for extra information.

At the time of screening A screening receptionist asks people who received the STI.VI. invitation (identified through a flag) whether they are interested in the STI.VI. study and therefore refers them to the STI.VI. desk.

At the STI.VI. desk, trained research assistants give further explanations and additional material (patient information sheet, informed consent form and the STI.VI. questionnaire). If informed consent is signed, an appointment is fixed for anthropometric measurements and for taking blood and saliva samples.

People are asked to fill in the questionnaire and to hand it back at the time of the blood sampling.

The STI.VI. questionnaire consists of 5 sections (physical activity, dietary habits, smoking habits, general health conditions, and general information) in order to collect baseline information on lifestyle habits. Type, amount and frequencies of dietary consumptions and physical activities are collected. The questionnaire also investigates the perception of one's own lifestyle and an motivation towards change.

In this study phase all participants are randomly allocated to the 4 study groups.

This is achieved through a permuted block design with block size of 12, 16, and 20 units width (W.F. Rosenberger, J. Lachin. Randomization in clinical trials: theory and practice. Wiley and sons, 2002, pag. 57). This method allows an almost complete uniform distribution of the randomisation groups in every moment of the study; this is necessary in order to simplify the subsequent courses management (see below). Participants are told about their group allocation at the time of biological sampling / anthropometric measurements, only.

At baseline appointment.

Participant subjects undergo anthropometric measurements. The following information are collected:

* Reproductive and eventual menopause history (women only)
* Eventual drug therapy under way,
* Height,
* Body composition,
* Waist circumference
* Arterial pressure. Then participants undergo blood drawing. Two types of blood samples are drawn: one for immediate biochemical analysis and another to be frozen. The freshly blood is used for instantaneous examinations for the following clinic-biochemical parameters: Insulin, Glucose, Total Cholesterol, LDL,HDL, Triglycerides, Minerals (Sodium, Potassium, Calcium, Iron), IGF-I, Testosterone, 17-ß-Estradiol, SHBG. These analyses are made for women invited to mammography screening while for people invited to colorectal screening supplemental tests are made also for vitamin D, 25 OH, PRC and high sensitive PRC.

Cryopreserved blood samples are stored in a bio-bank for epigenetic, metabolomics and metabonomics analyses. Bio-banking includes a security system and a data base specifically implemented for samples storage and traceability.

About 3 ml of saliva are also collected to investigate variations in genetic and metabolic parameters. Saliva samples are cryopreserved with the same modalities as blood samples.

Immediately after biological sampling / anthropometric measurements a short counselling takes place. Trained counsellors answer all eventual questions on the study posed by participants and inform them on the next steps. They also deliver to all participants a basic booklet containing general information on primary prevention, based on the most reliable and updated bibliographic sources on diet and physical exercise (World Cancer Research Fund/American Institute for Cancer Research. Food, nutrition, physical activity, and the prevention of cancer: a global perspective. Washington, DC: AICR, 2007; WHO, Move for Health, 2002; EU Working Group "Sport and Health", EU Physical Activity Guidelines, 2008).

Follow-up phase

Two follow-ups are planned:

• Intermediate, after 8 months since biological sampling / anthropometric measurements (the exact date is reckoned calculating 6 months + the average intervention duration ± 2 weeks, for managing reasons): it consists of repeating anthropometric measurements and questionnaire filling, and counselling.

All participants are contacted by letter and/or telephone, inviting them to contact the study secretariat in order to fix an appointment for repeating anthropometric measurements and questionnaire filling; during the follow-up visit trained counsellors verify participants' compliance with the provided recommendations, examine eventual encountered difficulties and provide support if needed.

• Final, after 6 months from intermediate follow-up (i.e., after 14 months since biological sampling / anthropometric measurements): it consists of repeating anthropometric measurements, biological sampling, and questionnaire filling, and counselling.

All participants are contacted by letter and/or telephone, inviting them to contact the study secretariat in order to fix an appointment for repeating once again anthropometric measurements, questionnaire filling and also biological sampling.

ELIGIBILITY:
Inclusion Criteria:

* 49 to 55-year-old women invited to mammography screening,
* 58 to 61 year-old people (both sexes) invited to colorectal screening

Exclusion Criteria:

* psychiatric disorders,
* disabling disease
* life expectancy <6 months
* eating or deambulation disorders
* in physiotherapy at the time of recruitment.

Ages: 49 Years to 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1270 (Actual)
Dates: Start 2010-05; Primary Completion 2014-01 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
feasibility outcome | 14 months
  initial participation rate overall and stratified by intervention group, age, and gender;
impact of intervention model | 14 months
  compliance to lifestyle recommendations and their maintenance assessed through the STI.VI. questionnaire;
impact of intervention model | 14 months
  changes in anthropometric measurements
impact of intervention model | 14 months
  comparison of metabolic parameters (insulin, glucose, total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides, IGF-1, testosterone)
impact of intervention model | 14 months
  evaluation of potential genetic and/or metabolic biomarkers in cancer development;
screening-related indicators | up to 10 years after study end
  screening participation rate in subjects enrolled in the STI.VI. study and, viceversa, STI.VI. participation rate in screened subjects;
screening-related indicators | up to 10 years after study end
  evaluation of breast and colorectal screening outcomes among STI.VI. participants

SECONDARY OUTCOMES:
Biobank implementation | up to 10 years after study end
  number of blood sample and saliva sample cryopreserved at baseline and at final follow up
Circulating biomarkers association with breast and colorectal cancer | up to 10 years after study end
  investigate whether selected circulating miRNAs previously found associated to brast and colorectal risk are significantly altered in the plasma of cancer patients compared to matched healthy controls and if they satisfy pre-specified true- and false positive rates that are considered minimally acceptable in the screening setting.

CONTACTS AND LOCATIONS:
Overall Officials: Nereo Segnan, MD MSc Epi, Principal Investigator — Director
Locations (1):
- S.C.D.O. Epidemiologia dei Tumori - Azienda Ospedaliera S. Giovanni Battista di Torino, Turin, Piedmont, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McBride CM, Emmons KM, Lipkus IM. Understanding the potential of teachable moments: the case of smoking cessation. Health Educ Res. 2003 Apr;18(2):156-70. doi: 10.1093/her/18.2.156. PMID 12729175
- [Background] Robb KA, Power E, Kralj-Hans I, Atkin WS, Wardle J. The impact of individually-tailored lifestyle advice in the colorectal cancer screening context: a randomised pilot study in North-West London. Prev Med. 2010 Dec;51(6):505-8. doi: 10.1016/j.ypmed.2010.10.002. Epub 2010 Oct 13. PMID 20950640
- [Background] Anderson AS, Mackison D, Boath C, Steele R. Promoting changes in diet and physical activity in breast and colorectal cancer screening settings: an unexplored opportunity for endorsing healthy behaviors. Cancer Prev Res (Phila). 2013 Mar;6(3):165-72. doi: 10.1158/1940-6207.CAPR-12-0385. Epub 2013 Jan 16. PMID 23324132
- [Background] Assfalg M, Bertini I, Colangiuli D, Luchinat C, Schafer H, Schutz B, Spraul M. Evidence of different metabolic phenotypes in humans. Proc Natl Acad Sci U S A. 2008 Feb 5;105(5):1420-4. doi: 10.1073/pnas.0705685105. Epub 2008 Jan 29. PMID 18230739
- [Background] Steindorf K, Ritte R, Eomois PP, Lukanova A, Tjonneland A, Johnsen NF, Overvad K, Ostergaard JN, Clavel-Chapelon F, Fournier A, Dossus L, Teucher B, Rohrmann S, Boeing H, Wientzek A, Trichopoulou A, Karapetyan T, Trichopoulos D, Masala G, Berrino F, Mattiello A, Tumino R, Ricceri F, Quiros JR, Travier N, Sanchez MJ, Navarro C, Ardanaz E, Amiano P, Bueno-de-Mesquita HB, van Duijnhoven F, Monninkhof E, May AM, Khaw KT, Wareham N, Key TJ, Travis RC, Borch KB, Sund M, Andersson A, Fedirko V, Rinaldi S, Romieu I, Wahrendorf J, Riboli E, Kaaks R. Physical activity and risk of breast cancer overall and by hormone receptor status: the European prospective investigation into cancer and nutrition. Int J Cancer. 2013 Apr 1;132(7):1667-78. doi: 10.1002/ijc.27778. Epub 2012 Sep 14. PMID 22903273
- See also: Related Info — http://apps.who.int/iris/bitstream/10665/67447/1/WHO_NMH_NPH_WHD_02.13.pdf